CLINICAL TRIAL: NCT01863992
Title: The Quality of Life a Direct Financial Costs Associated With Home Ventilation of Children: A Prospective Study
Brief Title: The Quality of Life and Direct Financial Costs Associated With Home Ventilation of Children: A Prospective Study
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Michael Seear, Principle Investigator, University of British Columbia
Other Study IDs: H13-00979
Record Dates: First submitted 2013-05-23; First posted 2013-05-29 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Children Receiving Ventilation at Home for Chronic Illness or Disease
Keywords: home ventilation
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators wish to learn about the quality of life (QOL) of children needing long term home ventilation and also that of their regular caregivers. In addition, the investigators will monitor the extra health-related expenses these families must meet. Data will be collected using two age-specific questionnaires of QOL plus a third one validated for assessing chronic health care costs. Questionnaires will be administered at an initial face to face meeting, supplemented by two telephone follow-up calls, to monitor medical expenses, one and two months later.

ELIGIBILITY:
Inclusion Criteria:

All families, or appointed guardians, caring for children that need home ventilatory support will be eligible for enrollment

Exclusion Criteria:

Refusal to join the study

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children receiving home ventilation for chronic illness or disease
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
The Quality of Life and Direct Financial Costs Associated With Home Ventilation | One year starting june 2013.
  Quality of life for children on home ventilation will be assessed using the validated PedsQL score. This has been specifically designed to measure quality outcome in children with long term health problems.

SECONDARY OUTCOMES:
The Quality of Life a Direct Financial Costs Associated With Home Ventilation | One year starting june 2013
  The quality of life for parents caring for a child needing home ventilation will be assessed using a validated questionnaire called the Caregiving Impact Scale (CIS)

OTHER OUTCOMES:
The Quality of Life and Direct Financial Costs Associated With Home Ventilation | One year starting june 2013
  The out-of-pocket expenses caused by caring for a child with home ventilation will be assessed using a validated questionnaire called the Ambulatory and Home Care Record (AHCR).

CONTACTS AND LOCATIONS:
Overall Officials: Mike Seear, MD, Principal Investigator — British Columbia's Children's Hospital; Mike Seear, MD, Principal Investigator — BCCH
Locations (1):
- BC's Children's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Seear M, Kapur A, Wensley D, Morrison K, Behroozi A. The quality of life of home-ventilated children and their primary caregivers plus the associated social and economic burdens: a prospective study. Arch Dis Child. 2016 Jul;101(7):620-7. doi: 10.1136/archdischild-2015-309796. Epub 2016 Mar 3. PMID 26940814